CLINICAL TRIAL: NCT01276249
Title: The STAPLE-International Post-Market Registry
Brief Title: The STAPLE International Post-Market Registry
Status: Terminated | Type: Observational
Why Stopped: Medtronic terminated the study since Foretevo product was no longer marketed
Sponsor: Medtronic Cardiovascular (Industry)
Responsible Party: Sponsor
Other Study IDs: CD03335-01
Record Dates: First submitted 2011-01-11; First posted 2011-01-13 (Estimated); Last update posted 2021-11-02 (Actual); Status verified 2021-10

CONDITIONS: Aortic Aneurysm, Abdominal; Aorto Iliac Aneurysm
Keywords: Aptus Endosystem; EndoStaple; Endograft; Stent Graft; Abdominal Aortic Aneurysm; Heli-FX; EndoAnchor
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Fortevo Endograft: All subjects diagnosed with a qualifying AAA suitable for elective endovascular repair, who meet the inclusion/exclusion criteria for the registry, are eligible for enrollment if treated with the Fortevo Endograft.
  Interventions: Device: Fortevo Endograft

INTERVENTIONS:
Device: Fortevo Endograft — The Fortevo Endograft, Main Body and Iliac Lumen Delivery System are indicated for the endovascular treatments of patients with infrarenal abdominal aortic aneurysms or aortic-iliac aneurysms having suitable morphology for endovascular repair.

SUMMARY:
The Aptus Endosystems STAPLE International Post-Market Registry is intended to expand the clinical knowledge base by including 'real world' subjects.

DETAILED DESCRIPTION:
The Aptus Endosystems STAPLE International Post-Market Registry is intended to expand the clinical knowledge base by including 'real world' subjects.

All subjects diagnosed with a qualifying AAA suitable for elective endovascular repair, who meet the inclusion/exclusion criteria for the registry, are eligible for enrollment and should be offered informed consent to participate.

ELIGIBILITY:
Inclusion Criteria:

1. Patient ≥ 18 years old
2. Patient has given written informed consent
3. Patient has a life expectancy > 1 year
4. Patient is willing to comply with follow-up evaluations
5. Patient's AAA meets at least one of the following criteria:

   * ≥ 4.5cm in diameter
   * Increased in size by 0.5cm in last 6 months
   * Maximum diameter exceeds 1.5 times the transverse dimension of an adjacent normal aortic segment
   * Saccular aneurysm larger than 3cm in maximal diameter
6. Patient has a proximal aortic neck diameter measured inner wall to inner wall between 19mm and 29mm
7. Patient has a proximal aortic neck length of at least 12mm
8. Patient has a patent iliac or femoral artery that allows endovascular access to the aneurysmal site with 16Fr (5.3mm) or 18Fr (6.0mm) delivery system.
9. Patient has bilateral iliac artery distal fixation site ≥ 10mm in length with an internal diameter between 9mm and 20mm

Exclusion Criteria:

1. Patient is participating in a concurrent clinical study which may confound STAPLE-International Registry results
2. Patient has a symptomatic AAA
3. Patient's AAA has a proximal aortic neck angle that is > 60 degrees between the infrarenal neck and the long axis of the aneurysm
4. Patient has irregularly-shaped plaque that would inhibit sealing stent apposition
5. Patient has aortic mural pathology that is ≥ 2mm in thickness over ≥ 50% of the circumference of the proximal fixation site
6. Patient has an active, or known history of, bleeding diathesis or hypercoagulable condition
7. Patient has a contraindication to any materials to which he or she will be exposed during the EVAR procedure (i.e., Fortevo Endograft or Heli-FX EndoAnchor System materials, contrast agents)
8. Patient has a genetic connective tissue disorder (e.g., Marfan's or Ehlers-Danloe Syndromes)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects diagnosed with a qualifying AAA suitable for elective endovascular repair.
Sampling Method: Non-Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2010-08; Primary Completion 2015-04 (Actual); Study Completion 2015-06-19 (Actual)

PRIMARY OUTCOMES:
Technical Success | Within 24 hours of the Index procedure
  The first primary endpoint is primary technical success. It consists of the following items:
  * Successful arterial access
  * Successful deployment of the Fortevo Endograft with secure proximal and distal fixation
  * Absence of type I or III endoleaks
  * Patent Fortevo Endograft without significant twist, kinking, or obstruction
Major Adverse Events (MAE) | Within 1-Month of Implantation
  The second primary endpoint is associated with the safety profile of the device, and is defined as the percent of patients experiencing one or more of major adverse events (MAE) within one month of implantation. MAE are defined as any one of the following events:
  * Death
  * Myocardial Infarction
  * Stroke (excludes TIA)
  * Renal failure (excludes renal insufficiency)
  * Respiratory Failure (excludes COPD or pulmonary complications)
  * Paralysis (excludes paraparesis)

SECONDARY OUTCOMES:
Clinical Success and Safety of the Fortevo Endograft and Heli-FX EndoAnchor System components | 1-Month, 6-Months and 12-Months
  Clinical Success is defined as Successful Deployment of the Fortevo Endograft at the intended location and the absence of:
  * Death as a result of aneurysm-related treatment
  * Type I or III endoleak
  * Fortevo Endograft infection
  * Fortevo Endograft thrombosis
  * Fortevo Endograft dilatation by 20% or more in diameter
  * Fortevo Endograft migration by 10mm or more at the proximal neck at 6-M and 12-M
  * Loss of Fortevo Endograft or Heli-FX EndoAnchor System integrity
  * Aneurysm expansion by 5mm (or more) in maximal diameter at 6-M and 12-M
  * Aneurysm rupture
  * Conversion to open repair

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Paul de Vries, MD, Principal Investigator — St Antonius Hospital - Nieuwegein, Netherlands
Locations (9):
- Sherbrooke University Hospital Centre, Sherbrooke, Quebec, Canada
- Germany (3):
  - German Heart Center, Berlin
  - Cardiovascular Center Frankfurt, Frankfurt
  - St. Bonifatious Hospital, Lingen
- Hellenic Airforce Hospital, Athens, Greece
- University of Siena, Siena, Italy
- St Antonious Hospital, Nieuwegein, Netherlands
- Spain (2):
  - Thorax Institute Hospital Clinic, Barcelona
  - University of Navarra, Pamplona

REFERENCES:
- [Background] Deaton DH. Future technologies to address the failed endoprosthesis. Semin Vasc Surg. 2009 Jun;22(2):111-8. doi: 10.1053/j.semvascsurg.2009.04.010. PMID 19573751
- [Result] Deaton DH, Mehta M, Kasirajan K, Chaikof E, Farber M, Glickman MH, Neville RF, Fairman RM. The phase I multicenter trial (STAPLE-1) of the Aptus endovascular repair system: results at 6 months and 1 year. J Vasc Surg. 2009 Apr;49(4):851-7; discussion 857-8. doi: 10.1016/j.jvs.2008.10.064. PMID 19341879